CLINICAL TRIAL: NCT07081321
Title: The Effect of Different Delivery Positions on Pelvic Floor Function.
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Gao lei, Attending Physician, Peking University People's Hospital
Other Study IDs: 2025PHB262-001
Record Dates: First submitted 2025-06-26; First posted 2025-07-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Stress Urinary Incontinence (SUI)
Keywords: Stress Urinary inconticence; Dlivery position; Pelvic Floor muscle strength
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lithotomy Position Group: Participants in the lithotomy position group were in the lithotomy position at the second stage of labor of delivery
  Interventions: Behavioral: Lithotomy position
- Upright Position Group: Participants in the upright position group were in the upright position at the second stage of labor of delivery.
  Interventions: Behavioral: Upright Position
- Lateral Position.: Participants in the lateral position group were in the lateral position at the second stage of labor of delivery.
  Interventions: Behavioral: Lateral Position

INTERVENTIONS:
Behavioral: Lithotomy position — Participants in the lithotomy decubitus position group were in the lithotomy position at the second stage of labor of delivery.
  Groups: Lithotomy Position Group
Behavioral: Lateral Position — Participants in the lateral position group were in the lateral position at the second stage of labor of delivery.
  Groups: Lateral Position.
Behavioral: Upright Position — Participants in the upright position group were in the upright position at the second stage of labor of delivery.
  Groups: Upright Position Group

SUMMARY:
This study is a cohort clinical study. Baseline data were collected from cases recruited at pregnancy, and the eligible subjects were grouped into 3 groups according to different delivery position including supine position group, upright position group, and lateral position group. Different delivery positions along with respectively timeand obstetric conditions were recorded at delivery. Pelvic floor function assessments were performed at postpartum.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-35 years old
2. Singleton, cephalic position, full-term primipara;
3. Cephalopelvic disproportion;
4. Expected fetal weight< 4000g;
5. Intended vaginal delivery in our hospital;
6. Voluntary participation of study subjects.

Exclusion Criteria:

1. Pelvic floor organ prolapse beyond the hymen limbus;
2. Combined with uncontrolled medical diseases and asthma, allergic rhinitis and constipation before pregnancy;
3. Presence of contraindications to vaginal delivery

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Singleton, cephalic position, full-term primipara aged 20-35 years old without cephalopelvic disproportion, expected fetal weight ≥ 4000gpelvic floor organ prolapse beyond the hymen limbus and combined with uncontrolled medical diseases and asthma, allergic rhinitis and constipation before pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 669 (Estimated)
Dates: Start 2025-12-07 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Stress urinary incontence (SUI) occurrence at 6 weeks postpartum | at 6 (±1) weeks postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Protection of research process and results
  • For unpublished research, data sharing may lead to the results being published first, damaging the academic rights and interests of the research team.